CLINICAL TRIAL: NCT02978586
Title: A Pilot Study of [Ga-68]PSMA PET/MRI for the Assessment of PSMA-positive Tumors
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE7Y16
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Prostate-specific Membrane Antigen Positive Tumors; Prostate Cancer; Breast Cancer; Lung Cancer
Keywords: PSMA; PET/MRI
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- [Ga-68]PSMA PET/MR: Up to 3 experimental PET/MRI scans will be performed to determine the level of [Ga-68]PSMA tumor uptake
  Interventions: Device: [Ga-68]PSMA PET/MR

INTERVENTIONS:
Device: [Ga-68]PSMA PET/MR — All participants will undergo at least 1 baseline [Ga-68]PSMA PET/MR. If participants test positive for [Ga-68]PSMA tumor uptake, they will under up to 2 additional scans
  Other Names: PET/MRI

SUMMARY:
The purpose of this study is to see if positron emission tomography/ magnetic resonance imaging (PET/MRI) can be used to monitor the effectiveness of cancer treatment using an investigational radioactive drug called [Ga-68]PSMA.

DETAILED DESCRIPTION:
Primary Objective

The primary objective of this pilot imaging study is to determine the feasibility of using positron emission tomography/ magnetic resonance (PET/MR) with [Ga-68] prostate-specific membrane antigen (PSMA) for staging and treatment monitoring of PSMA expressing tumors. [Ga-68]PSMA PET/MR findings will be compared with standard of care imaging, patient follow up, and histopathology if available. [Ga-68]PSMA PET/MR will not be used to change the patients' treatment plan. Investigators will assess PET/MR test-retest reproducibility and compare baseline [Ga-68]PSMA PET/MR with PET/MR after initiation (within 2-6 weeks) of therapy and evaluate if [Ga-68]PSMA is a suitable biomarker for treatment monitoring and assessment of early treatment response.

Secondary Objectives

* To compare early changes in PET biomarker ([Ga-68]PSMA) tumor uptake with treatment response assessed at completion of therapy (prediction of treatment response).
* To compare changes in MRI signal intensities (multi-parametric MRI) with treatment response assessed at completion of therapy.
* To compare results from multi-parametric MR imaging with [Ga-68]PSMA uptake.
* To assess combinations of quantitative PET and MRI metrics.

Study Design Patients, who enroll in this study, will undergo a baseline [Ga-68]PSMA PET/MR to assess the level of [Ga-68]PSMA tumor uptake. Patients with positive [Ga-68]PSMA tumor uptake (defined as [Ga-68]PSMA uptake twice the background activity) who are receiving systemic therapy will undergo a further [Ga-68]PSMA PET/MR 2-6 weeks after start of treatment. Patients with positive [Ga-68]PSMA tumor uptake will also be offered to participate in a test- retest study with a 2nd [Ga-68]PSMA PET/MR prior to treatment. Patients will therefore undergo a maximum of three [Ga-68]PSMA PET/MR imaging procedures. The first two test-retest Ga-PSMA-PET/MRI will be performed on separate days to allow for radioactive decay. There will be no other (e.g. clinically indicated) PET scan performed on the same day of [Ga-68]PSMA-PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PSMA-positive tumors including prostate cancer, breast cancer, lung cancer, and other tumor types know to express PSMA
* Patients able to tolerate PET/MRI scans
* Informed consent must be given and signed

Exclusion Criteria:

* Subjects who do not meet the above mentioned inclusion criteria
* Subjects who refuse to give and/or sign the informed consent
* Patients who have a history of serious adverse events related to a previous MRI or PET/CT
* Patients who are unable to undergo MRI scanning due to exclusion by institutional MRI restriction policies as mentioned in the standard institutional MRI informed consent form
* Patients who are currently pregnant or breast feeding. A pregnancy test within 72 hours of the first PET/MRI will be performed.
* Anti-cancer treatment (chemotherapy and/or radiation therapy) within the last 2 weeks.
* Renal insufficiency: elevated Creatinine and/or Glomerular Filtration Rate (GFR)<40ml/min/1.7sqm (exclusion criterion only for contrast enhanced MRI)
* Patients with a known allergy against any component of the contrast enhancing MR agent will not receive MR contrast agents. (exclusion criterion only for contrast enhanced MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with tumors expressing PSMA including prostate cancer, breast cancer, lung cancer, renal cancer and other tumor types [Ga-68]PSMA PET/MRI known to express PSMA
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Test-retest reproducibility of PET biomarker ([Ga68]-PSMA) uptake using PET/MRI | Up to 6 weeks after beginning treatment
  The outcome measure for the statistical analysis of the test-retest reproducibility will be concordance analysis of standard uptake values (SUVs) between the 2 baseline scans

SECONDARY OUTCOMES:
Test-retest reproducibility of quantification of MRI sequences (multi-parametric MRI) | Up to 6 weeks after beginning treatment
  Morphologic imaging will be performed based on standard of care imaging protocols for anatomic detail and localization. Quantitative analysis will include Diffusion weighted imaging (DWI) and Dynamic contrast enhanced MRI (DCE-MRI)
Ability of PET/MRI to measure changes in PET biomarker [Ga-68]PSMA) tumor uptake after initiation of therapy | Up to 6 weeks after beginning treatment
  A region of interest (ROI) will be placed in tumor lesions on the digital PET images in order to obtain Standardized Uptake Values (SUV) and/or time activity curves (TACs).
  Relative and absolute differences in tumor SUVs between pre-treatment PET vs. PET after initiation of therapy will be calculated. These differences in [Ga-68]PSMA tumor uptake will be compared with treatment response at completion of therapy (prediction of treatment response).
Changes in MR signal intensities after initiation of therapy | Up to 6 weeks after beginning treatment
  Standard morphologic imaging will be obtained in a target area harboring tumor tissue before and after treatment. Quantitative parameters will be obtained in the respective techniques by drawing a region of interest (ROI) in the tumor lesions using dedicated post processing software and interactive workstations. Relative and absolute differences in tumor signal intensities and quantitative parameters will be calculated between pre-treatment PET vs. PET after initiation of therapy. These differences will be compared with treatment response at completion of therapy (prediction of treatment response) as assessed by standard of care imaging
Comparison of early changes in PET biomarker ([Ga68]PSMA) tumor uptake with treatment response assessed at completion of therapy | Up to 6 weeks after beginning treatment
  Relative and absolute differences in tumor SUVs between pre-treatment PET vs. PET after initiation of therapy will be compared with treatment response at completion of therapy.
Comparison of changes in MRI signal intensities (multi-parametric MRI) with treatment response assessed at completion of therapy | Up to 6 weeks after beginning treatment
  Relative and absolute differences in tumor MRI signal intensities and quantitative parameters as described above between pre-treatment PET vs. PET after initiation of therapy will be compared with treatment response at completion of therapy.
Comparison of results from multi-parametric MR imaging with [Ga-68]PSMA tumor uptake | Up to 6 weeks after beginning treatment
  Changes of tumor Ga68-PSMA uptake between baseline and during treatment will be compared with changes in MR multiparametric imaging (e.g. apparent diffusion coefficient (ADC) maps, MR perfusion parameters, changes in T2* maps, etc.). The ability of each PET and MR parameter will be assessed for the ability to predict treatment response.
Assessment of combinations of quantitative PET and MRI metrics | Up to 6 weeks after beginning treatment
  Investigators will assess combinations of quantitative PET and MRI metrics regarding their ability to characterize tumors and predict treatment response. Advanced feature extraction and pattern recognition methods will be used to find a combination of fused MRI and PET features that are correlated with disease signature.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Avril, MD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals, Case Comprehensive Cancer Center, Cleveland, Ohio, United States